CLINICAL TRIAL: NCT02910531
Title: The Effect of Lipoic Acid Natural Supplement on Cystine Stone Formation
Brief Title: Lipoic Acid Supplement for Cystine Stone
Acronym: ALA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Chi, MD (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Thomas Chi, MD, Professor, Urology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16-20523; 2P20DK100863-03 (NIH); OPD Grant Number 5716 (Other Grant/Funding Number: US Food and Drug Administration)
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Cystinuria
Keywords: Cystinuria; Kidney stone; Alpha lipoic acid
MeSH Terms: conditions — Cystinuria; Kidney Calculi | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALA supplement (Experimental): Clinical data including medical history, plain KUB x-ray and renal ultrasound, routine blood work and 24-hour urine collections for all subjects will be collected as part of normal clinical care at routine clinical visit every 4 months.
  Subjects in this study arm will be taking one supplement tablet containing 1200 mg of alpha lipoic acid orally once daily for three years.
  At the end of the three years of study drug treatment, all subjects will undergo a low dose non-contrast CT scan to look for a silent change in stone size.
  Interventions: Dietary Supplement: Alpha lipoic acid
- Placebo (Placebo Comparator): Clinical data including medical history, plain KUB x-ray and renal ultrasound, routine blood work and 24-hour urine collections for all subjects will be collected as part of normal clinical care at routine clinical visit every 4 months.
  Subjects in this study arm will be taking one placebo tablet containing 10 mg of sucrose orally once daily for three years.
  At the end of the three years of study drug treatment, all subjects will undergo a low dose non-contrast CT scan to look for a silent change in stone size.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Alpha lipoic acid — Already mentioned in arm/group descriptions.
  Arms: ALA supplement
Drug: Placebo — Already mentioned in arm/group descriptions.
  Arms: Placebo

SUMMARY:
This study evaluates how daily alpha lipoic acid supplementation affects cystine kidney stone recurrence. Half of the subjects will receive 1200 mg alpha lipoic acid orally daily for three years, while the other half will receive a placebo. The funding source for this clinical trial is FDA OOPD.

DETAILED DESCRIPTION:
Cystinuria is a rare inherited autosomal recessive disorder of the kidney that is the result of a defect in the dibasic amino acid transporter in the renal proximal tubule and small intestine. Supersaturation of cystine in the urine produces crystals that precipitate and form calculi, which can be a cause of obstruction, infection, and chronic kidney disease (Chillarón 2010).

One potential therapeutic is a thiol-containing compound alpha-lipoic acid (thioctic acid, 5-(1,2-dithiolan-3- yl) pentanoic acid, ALA). It is an over-the-counter supplement with antioxidant property. Once ALA is transported into the cell, it is reduced to dihydrolipoic acid (DHLA). Both ALA and DHLA have direct antioxidant activity (Scholich 1989), and they can regenerate endogenous antioxidants including ascorbic acid and vitamin E. It can also increase intracellular coenzyme Q10 and glutathione levels. ALA and DHLA also have additional biochemical effects as metal chelators, reactive oxygen species scavengers, and modulators of signaling transduction of several pathways (Gomes 2014).

While the potential therapeutic effects of ALA have been studied in a number of diseases including, for example, Alzheimer's disease, obesity, cardiovascular disease, hypertension, and several cancers (Gomes 2014), the efficacy of ALA has been best studied in type 2 diabetic peripheral neuropathy (Ziegler 2011). In our lab, results from a mouse model of cystinuria show that ALA markedly slows the initiation of cystine stone formation as well as the growth of existing stones.

Given this history in clinical medicine and, most importantly, based upon our positive findings of ALA effectiveness in a mouse model of cystinuria, we propose a pilot study on the use of this molecule in cystinuric patients.

ELIGIBILITY:
Inclusion Criteria:

* Documented cystinuria on prior 24-hour urine collection and/or stone analysis; history of previous cystine kidney stones.
* Being able and willing to provide consent.

Exclusion Criteria:

* Poorly controlled diabetes mellitus (hemoglobin A1C > 8.0% for more than 1 year).
* Current alpha-lipoic acid administration at the time of screening or within the last year prior to screening.
* Vulnerable populations including incarceration status.
* Unable to give informed consent.
* Non-English primary language.
* Pregnancy, lactation, or child-bearing age without birth control devices.
* Anticipation of pregnancy during the study period.
* Serious illness likely to cause death within the next 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Cystine stone recurrence | 3 years
  The primary efficacy endpoint will be assessed in two ways:
  1. symptomatic stone recurrences, defined as renal colic, stone passage, or surgical removal of a stone;
  2. silent stone recurrences, classified as stone growth or new stones, diagnosed on the basis of renal ultrasound, plain KUB x-ray, or if clinically indicated, computed tomography.

SECONDARY OUTCOMES:
Urinary cystine level | 3 years
  The secondary endpoints will be quantitative urinary cystine level determined by 24-hour urine collection.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chi, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chillaron J, Font-Llitjos M, Fort J, Zorzano A, Goldfarb DS, Nunes V, Palacin M. Pathophysiology and treatment of cystinuria. Nat Rev Nephrol. 2010 Jul;6(7):424-34. doi: 10.1038/nrneph.2010.69. Epub 2010 Jun 1. PMID 20517292
- [Background] Gomes MB, Negrato CA. Alpha-lipoic acid as a pleiotropic compound with potential therapeutic use in diabetes and other chronic diseases. Diabetol Metab Syndr. 2014 Jul 28;6(1):80. doi: 10.1186/1758-5996-6-80. eCollection 2014. PMID 25104975
- [Background] Ziegler D, Low PA, Litchy WJ, Boulton AJ, Vinik AI, Freeman R, Samigullin R, Tritschler H, Munzel U, Maus J, Schutte K, Dyck PJ. Efficacy and safety of antioxidant treatment with alpha-lipoic acid over 4 years in diabetic polyneuropathy: the NATHAN 1 trial. Diabetes Care. 2011 Sep;34(9):2054-60. doi: 10.2337/dc11-0503. Epub 2011 Jul 20. PMID 21775755
- [Background] Scholich H, Murphy ME, Sies H. Antioxidant activity of dihydrolipoate against microsomal lipid peroxidation and its dependence on alpha-tocopherol. Biochim Biophys Acta. 1989 Feb 20;1001(3):256-61. doi: 10.1016/0005-2760(89)90108-2. PMID 2492825